CLINICAL TRIAL: NCT00085657
Title: Enhancement of Rehabilitative Treatment-Dependent Functional Recovery After Stroke by Transcranial Direct Current Stimulation (tDCS)
Brief Title: Brain Electrical Stimulation to Enhance Recovery After Stroke
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040212; 04-N-0212
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-05-21

CONDITIONS: Stroke
Keywords: Direct Current Stimulation; Cortical Reorganization; Rehabilitation; Acute Stroke; Stroke
MeSH Terms: conditions — Stroke

SUMMARY:
This study will examine whether brain stimulation using transcranial direct current stimulation (tDCS) in stroke patients undergoing rehabilitation therapy can help patients recover strength and motor function more than rehabilitation therapy alone. For tDCS, two small metal disks (electrodes) attached to wires are placed on small cotton pads and taped to the subject's head, one on the forehead above the eye and the other on the top of the head. The electrodes deliver a brief electrical current that stimulates the cortex, the part of the brain responsible for motor function.

Adult patients who have weakness on one side of their body as a result of a stroke occurred within the last 15 days may be eligible for this study. NIH is not directly recruiting patients for this study. Patients will be selected through the National Rehabilitation Hospital (NRH) Research Center personnel in Washington, DC, from patients under treatment at that facilitiy. Candidates are screened with a physical and neurologic examination, a review of tests done on admission to NRH, and a magnetic resonance imaging (MRI) scan, if one has not been done since the stroke. MRI uses a strong magnetic field and radio waves to obtain images of the brain. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, the patient lies on a table that can slide in and out of the cylinder. Scanning time for this study takes about 30 to 45 minutes.

Participants are randomly assigned to receive tDCS or placebo stimulation, along with rehabilitation therapy, for 2 to 3 weeks, depending on the patient's length of stay at the NRH. For the placebo stimulation, electrodes are placed on the patient's scalp as with tDCS, but no current is delivered. Before and after each rehabilitation session with electrodes, patients undergo Jebsen Taylor motor testing, in which they are asked to lift small objects, turn cards, use a spoon, stack checkers, and lift cans as fast as they can.

On the day of discharge, patients have physical and neurological examinations and the motor function tests described below. The motor tests are repeated, along with standard care and a review of their health status, during outpatient follow-up visits scheduled at 3, and 12 months. The motor tests are:

* Wolf motor function test - Patients are asked to raise a forearm on a table, on a box, to reach across a table, push a sandbag, place a hand on the table, pull a weight, lift a can, pick up a pencil, pick up a paper clip, stack checkers, flip cards, use a key, fold a towel, and pick up a basket.
* Barthel index - Patients are timed for the speed with which they perform certain tasks, such as feeding, grooming, or moving a wheelchair.
* Abilhand questionnaire - Patients answer questions about how they perform routine daily activities.
* GOT test of tactile discrimination - Patients describe objects they feel with their hand.
* Ashworth spasticity scale - A medical staff person moves the patient's arm back and forth to see how stiff it is.

DETAILED DESCRIPTION:
OBJECTIVES

There is no universally accepted strategy to promote recovery of motor function after stroke, the main cause of long-term disability among adults. Neurorehabilitation contributes to recovery during the first days to weeks after stroke and later decelerates. Therefore, it is desirable to develop strategies to enhance rehabilitative effects on motor recovery particularly in the early phase after stroke in this patient group. We have recently demonstrated that cortical stimulation in the form of TMS enhances the beneficial effects of motor training and cortical plasticity in healthy volunteers and that tDCS (another noninvasive more comfortable stimulating technique than TMS transiently improves functional motor skills of the paretic hand of chronic stroke patients in the absence of training. Given the paucity of strategies available to enhance neurorehabilitation after stroke, it is now crucial to determine if tDCS can enhance the beneficial effects of customarily used rehabilitative treatment. tDCS has been used in several hundred subjects worldwide and in approximately 9 stroke patients, 15 Parkinson's disease patients and 15 healthy volunteers in our lab in the absence of undesirable side effects.

In addition to the above objectives, we will also apply functional magnetic resonance imaging (fMRI) and transcranial magnetic stimulation (TMS) techniques to determine the extent of changes in neural responses and functional shift in cortical representations/reorganization as a result of the proposed intervention strategies. fMRI as a measure is important in understanding changes in brain activation prior to, during, and after motor recovery and the effects of tDCS and the rehabilitative treatment strategies under investigation. Integrating TMS together with fMRI studies will provide crucial information on the functional role of brain regions activated in neuroimaging studies in association with functional recovery.

STUDY POPULATION

We plan to study 120 patients with a single cortical or subcortical subacute stroke. Thirty healthy volunteers and a sub-group of 30 patients from the 120 patient population will also be recruited in the fMRI and TMS part of the study. The reason for including 30 patients in the fMRI and TMS components of the study is that it is anticipated that not all the 120 patients recruited in the initial study (i.e., the tDCS and therapeutic intervention phase) may be able to perform the tasks required for the fMRI part of the study and also satisfy the Exclusion criteria for fMRI scans. In addition, based on previous studies and preliminary fMRI power analysis, we estimate that 30 patients is likely to be sufficient to provide a representative sample of the patient group for the testing of the hypotheses stated in the protocol. Thirty healthy volunteers are necessary for the fMRI and TMS components of the study in order to obtain normative data for the TMS and fMRI components of the investigation. They will have the multiple number of TMS and fMRI sessions as patients in order to obtain descriptive information on the variability of these measures in both groups.

DESIGN

The purpose of this protocol is to test the hypothesis that tDCS applied in combination with customary rehabilitative training as used in the community (RT) will enhance motor recovery 3 months after admission relative to placebo and RT, and that functional recovery is associated with changes in cortical excitability in the ipsilesional primary motor cortex (M1) and dorsal pre-motor cortex. The tDCS part of the study will be done at the NRH (where is being evaluated in parallel with the NINDS review process). Patients will be included in the protocol as soon as they are admitted to the NRH for RT (usually 3-10 days after the ictal event). Patients, who are eligible for the protocol will be randomized in one of the two study arms: RT + tDCS or RT + placebo stimulation. In both study arms patients will take part in daily customary RT procedures. We will record the specific rehabilitative therapy received by the patient. In the tDCS study arm, patients will receive tDCS of the motor cortex associated with RT every other day for the time of the inpatient stay (14 days). Placebo will be implemented in the same way and with the same stimulating equipment in place as tDCS. Patient and therapist (who will provide treatment and determine the primary outcome measure) will not be aware of arm participation (double-blind study design).

Normal volunteers will be recruited only for the fMRI and TMS part of the study which will be carried out at the NIH. They will be screened based on the criteria listed in the protocol and receive a neurological exam to determine their qualification for the proposed studies.

OUTCOME MEASURES

Primary outcome measure will be the Jebsen-Tailor-Test (JTT), a test measuring the functional abilities of the hand in daily living activities. Secondary outcome measures will include the Wolf Motor Function Test (WMFT), the Fugl-Meyer-scale (FMS), the MRC scale, the Abilhand scale (AHS), Barthel Index, Ashworth-Spasticity scale (ASS), and grating orientation task (GOT) and the NIH stroke scale. For the fMRI and TMS studies, changes in BOLD (blood oxygenation level dependent) response and delayed reaction time will be the outcome measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include patients aged 18-80 years old with subacute thromboembolic non-hemorrhagic subcortical or cortical strokes stratified according to the degree of impairment into mildly impaired (MRC greater than 3) and severely impaired (MRC less than 3). Assessment of the initial functional state will be taken at the admission at NRH. For healthy volunteers, subjects with a normal physical and neurological examination could participate.

EXCLUSION CRITERIA:

1. Patients with more than one stroke in the medial cerebral artery territory.
2. Patients with bilateral motor impairment.
3. Patients with cerebellar or brainstem lesions.
4. Patients with history of severe alcohol or drug abuse, psychiatric illnesses like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 23 or less).
5. Patients with severe uncontrolled medical problems (e.g. cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others).
6. Patients with increased intracranial pressure as evaluated by clinical means.
7. Patients with unstable cardiac arrhythmia.
8. Patients with thyroid disorders.
9. Patients with more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease.
10. Pregnancy.
11. Patients with metallic implants in the head.
12. Patients with pacemakers.
13. Patients taking antiadrenergic medications.
14. For fMRI: 1) Medical or technical contraindications to MRI procedures (e.g. metal braces, pacemakers, cochlear devices, surgical clips, and other metal/magnetic implants); 2) Claustrophobia; 3) inability to comply with the protocol 4) pregnancy (a urine pregnancy test will be performed for premenopausal females prior to MRI). All other criteria stated above will also apply
15. For TMS: 1) Seizure disorder; 2) Metallic implant in the head; 3) Pacemaker; 4) Unable to perform the task; 5) Pregnant or breast feeding a child; 6) Patients or subjects with increased intracranial pressure as evaluated by clinical means. All other criteria stated above will also apply.

For healthy volunteers, subjects with stroke(s) or movement disorder(s); history of alcohol or drug abuse or a psychiatric illness like depression, other major medical problems that effect heart, lungs or kidneys or epilepsy or diabetes mellitus; thyroid gland problem; other diseases of the brain, like Alzheimer's disease; medical or technical contraindications to MRI procedures (e.g. metal braces, pacemakers, cochlear devices, surgical clips, and other metal/magnetic implants); claustrophobia; pregnant or breast feeding women could not participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-06-09; Study Completion 2009-05-21

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Rehabilitation Hospital Research Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Background] Hackel ME, Wolfe GA, Bang SM, Canfield JS. Changes in hand function in the aging adult as determined by the Jebsen Test of Hand Function. Phys Ther. 1992 May;72(5):373-7. doi: 10.1093/ptj/72.5.373. PMID 1631206
- [Derived] Hodics TM, Nakatsuka K, Upreti B, Alex A, Smith PS, Pezzullo JC. Wolf Motor Function Test for characterizing moderate to severe hemiparesis in stroke patients. Arch Phys Med Rehabil. 2012 Nov;93(11):1963-7. doi: 10.1016/j.apmr.2012.05.002. Epub 2012 May 10. PMID 22579647